CLINICAL TRIAL: NCT07233018
Title: A Clinical Study to Investigate the Safety and Efficacy of CT0991 in Patients With Relapsed/Refractory Acute Myeloid Leukemia.
Brief Title: A Clinical Study to Explore the Safety and Efficacy of CT0991 in Relapsed/ Refractory Acute Myeloid Leukemia
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: MEI HENG (Other)
Responsible Party: Sponsor-Investigator, MEI HENG, Principal Investigator, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Organization: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CT0991-CG9001_01
Record Dates: First submitted 2025-11-13; First posted 2025-11-18 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Relapsed/Refractory Acute Myeloid Leukemia(AML)
Keywords: CT0991
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CAR-T cells# chimeric antigen receptor T cells# (Experimental): CT0991 CAR-T cels inffusicn
  Interventions: Drug: CT0991 CAR-T cells infusicn

INTERVENTIONS:
Drug: CT0991 CAR-T cells infusicn — CAR-T cells# chimeric antigen receptor T cells#

SUMMARY:
A Clinical Study to Investigate the Safety and Efficacy of CT0991 in Patients with Relapsed/Refractory Acute Myeloid Leukemia.

DETAILED DESCRIPTION:
This is a single-arm, open-label, dose-escalation clinical trial to evaluate the safety, efficacy, and cellular pharmacokinetics of CT0991 in patients with relapsed or refractory acute myeloid leukemia. It is planned to enroll 3-24 participants in this trial.

ELIGIBILITY:
Inclusion Criteria:

1. Volunteer to participate in the clinical trial; Fully understand and are informed of this study and sign the informed consent form; Willing to follow and able to complete all trial procedures.
2. Age 18-75 years (inclusive), male or female.
3. Estimated survival > 12 weeks.
4. Patients with relapsed or refractory AML as defined in the Chinese Guidelines for the Diagnosis and Treatment of Relapsed and Refractory Acute Myeloid Leukemia (Version 2023);
5. Flow cytometry or immunohistochemical examination of bone marrow or peripheral blood samples showed positive expression of CD38 in tumor cells and the expression rate was ≥80%.
6. ECOG score 0-2.
7. Participants should meet the following test results (no ongoing supportive care):

   1. Left ventricular ejection fraction (LVEF) > 50%;
   2. ALT≤ 2.5 × ULN, AST ≤ 2.5 × ULN, total bilirubin ≤ 2 × ULN;
   3. Endogenous creatinine clearance ≥ 30 mL/min (creatinine clearance calculated using the Cockcroft-Gault formula);
   4. Activated partial thromboplastin time (APTT) ≤ 1.5 × ULN and prothrombin time (PT) ≤ 1.5 × ULN.

Exclusion Criteria:

1. The participant has any serious illness, laboratory abnormality, or psychiatric disorder that may impair the ability to receive or tolerate planned trial treatment; or the investigator judges that the participant's participation in the clinical trial is not in his/her best interest (e.g.,compromised health), or may hinder, limit, or confound protocol-specific Assessments.
2. Participants were diagnosed with acute promyelocytic leukemia (APL),BCR-ABL positive leukemia (chronic myeloid leukemia in acute phase),secondary AML (other than MDS), central nervous system leukemia.
3. Participants with a history of epilepsy or other central nervous system disease;
4. Participants who have previously received autologous or allogeneic CAR-T therapy.
5. Participants who have received autologous stem cell transplantation or allogeneic stem cell transplantation within 12 weeks.
6. Participants who have received prior immunotherapy targeting CD38.
7. Participant has clinically significant active GVHD or is receiving systemic corticosteroids for GVHD.
8. Participant has any of the following at screening:

1)Active, uncontrolled systemic infection or requiring intravenous anti-infective agents.

2)Any of the following cardiac conditions, including:

1. New York Heart Association Class III-IV heart failure;
2. History of myocardial infarction, coronary artery bypass grafting, or unstable angina within 6 months prior to Qinglin;
3. History of uncontrolled arrhythmia of significant clinical significance (as judged by the investigator), such as ventricular arrhythmia;
4. History of severe nonischemic ardiomyopathy;
5. Other cardiac disease that the investigatorbelieve could jeopardize the participant 's well-being or compromise participation in this clinical trial; 3) Active bleeding of clinical significance as judged by the investigator; 4)Requiring supplemental oxygen to maintain oxygen saturation> 92%; 5)Patients with severe chronic obstructive pulmonary disease (COPD) or other lung diseases that cannot tolerate CAR-T treatment as judged by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-11-18 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2027-05-30 (Estimated)

PRIMARY OUTCOMES:
MTD and/or dose range | Up to 28 days after CAR-T cells infusion
  Evaluate Dose limited toxicity and recommended dosage range after CT0991 infusion.
Adverse Events (AE) after CT0991 infusion | 12 months after CT0991 infusion
  An assessment of severity grade will be made according to the National Cancer Institute Common Terminology Criteria.
Dose-limiting toxicity （DLT） | Up to 28 days after CAR-T cells infusion.
  The DLT is evaluated as the proportion of patients who experienced adverse events related to CT0991 that meet the criteria for DLT events after the first infusion.

SECONDARY OUTCOMES:
Complete response (CR), complete response with partial hematologic recovery (CRh) | 12 months after CT0991 infusion.
  and complete response with incomplete hematologic recovery (CRi).Performed according to the Technical Guidelines for Clinical Development of New Drugs for Acute Myeloid Leukemia and ELN 2022 Criteria for AML defined of Achieve CR、CRh and CRi.
Morphologic leukemia-free status (MLFS) and partial response (PR) | 12 months after CT0991 infusion
  Performed according to the Technical Guidelines for Clinical Development of New Drugs for Acute Myeloid Leukemia and ELN 2022 Criteria for AML defined of Achieve CRh, MLFS and PR.
Duration of response （DOR) | 12 months after CT0991 infusion.
  Participants achieving CR/CRi/CRh will be included in the analysis set for DOR. DOR is defined as the time from the date of confirmed response until the date of disease relapse or death from any cause, whichever occurs first.
Event-free survival (EFS) | 12 months after CT0991 infusion.
  Defined as the time from the date of receiving the infusion to the date of treatment failure (failure to achieve CR/CRh/CRi/MLFS/PR after both efficacy assessments), or relapse (hematologic relapse or extramedullary relapse after CR/CRh/CRi), or death from any cause, whichever occurs first. When an EFS event was "Ineffective Therapy", the primary analysis of EFS was performed on a 1-day basis (ie, time to treatment received as the event). For a more comprehensive assessment, sensitivity analyses could be performed using the actual date of treatment failure, end of treatment, or start of next-line anti-leukemia therapy as the end of EFS for treatment failure, respectively.
Overall survival (OS) | 12 months after CT0991 infusion.
  Defined as the time from the date of receiving the infusion to the date of death from any cause.
Minimal Residual Disease (MRD) Negative Rate | 12 months after CT0991 infusion.
  tested in all participants who achieved CR/CRh/CRi. MRD negativity was defined as abnormal cells detected by the MFC method accounting for < 0.1% of CD45-positive cells.
Pharmacokinetic parameters of CT0991, including CAR copy number, peak value, AUC (area under the curve), in vivo persistence, etc. | 12 months after CT0991 infusion.
  Time to peak expansion, peak expansion, area under the curve (AUC) and duration in plasma after infusion of CT0991 cells.

CONTACTS AND LOCATIONS:
Locations (1):
- Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No